CLINICAL TRIAL: NCT00001906
Title: Safety and Immunogenicity of a Vaccine for Cutaneous Leishmaniasis Using Recombinant Human Interleukin-12 and Aluminum Hydroxide Gel as Adjuvants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 990091; 99-I-0091
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-04

CONDITIONS: Cutaneous Leishmaniasis
Keywords: Alum; Antigen; Cytokine; Parasitic Infection; Phase I; Cutaneous Leishmaniasis
MeSH Terms: conditions — Leishmaniasis, Cutaneous; Parasitic Diseases | interventions — Interleukin-12

INTERVENTIONS:
Biological: Combination of autoclaved leishmania antigen with recombinant human interleukin-12 (rhIL-12) and aluminum hydroxide gel as adjuvants

SUMMARY:
While vaccination against cutaneous leishmaniasis, a chronic ulcerating protozoan infection of the skin, has been possible for decades using live parasites, the production and storage of live cultures are difficult. Since inoculation occasionally leads to severe infection, most experts now advocate against their use. We have shown excellent protection using a "heat-killed" vaccine that combines autoclaved leishmania antigen with recombinant human interleukin-12 (rhIL-12) and aluminum hydroxide gel as adjuvants in a rhesus macaque model of disease. To assess the safety and immunogenicity of this vaccine in humans, we now propose a rhIL-12 dose escalation Phase I/II trial.

DETAILED DESCRIPTION:
While vaccination against cutaneous leishmaniasis, a chronic ulcerating protozoan infection of the skin, has been possible for decades using live parasites, the production and storage of live cultures are difficult. Since inoculation occasionally leads to severe infection, most experts now advocate against their use. We have shown excellent protection using a "heat-killed" vaccine that combines autoclaved leishmania antigen with recombinant human interleukin-12 (rhIL-12) and aluminum hydroxide gel as adjuvants in a rhesus macaque model of disease. To assess the safety and immunogenicity of this vaccine in humans, we now propose a rhIL-12 dose escalation Phase I/II trial.

ELIGIBILITY:
Male or non-pregnant female 18 - 50 years of age at the time of screening and willing to use effective birth control for one month post vaccination.

Free of obvious health problems as established by medical history and clinical examination before entering into the study.

Available to participate for the duration of the study (approximately 6 months).

Able to give signed informed consent.

May not have received an investigational leishmania vaccine or skin test, or recombinant human interleukin-12.

No use of an investigational drug or any vaccine other than the study vaccine within 30 days preceding the dose, or planned use during the study period.

No administration of chronic immunosuppressants (defined as more than 14 days) or other immune-modifying drugs within six months of vaccination. (For corticosteroids, this will mean prednisone, or equivalent, greater than 0.5 mg/kg/day. Inhaled and topical steroids are allowed.)

No history of prior leishmaniasis or of extensive travel to regions endemic for leishmaniasis, such as southern Mexico, Central and most of South America, the Mediterranean region and Middle East, Africa, and India.

No confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.

No family history of congenital or hereditary immunodeficiency.

No history of significant allergic disease or reactions likely to be exacerbated by any component.

No acute disease at the time of enrollment, defined as the presence of a moderate or severe illness with or without fever.

No acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal function abnormality, as determined by physical examination or laboratory screening tests.

No pregnant or lactating females.

Must not have suspected or known alcohol or drug abuse.

No other significant finding that, in the opinion of the investigator, would increase the risk of having an adverse outcome from participating in this study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 1999-04; Study Completion 2001-05

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Guirges SY. Natural and experimental re-infection of man with Oriental sore. Ann Trop Med Parasitol. 1971 Jun;65(2):197-205. doi: 10.1080/00034983.1971.11686746. No abstract available. PMID 4253634
- [Background] Naggan L, Gunders AE, Michaeli D. Follow-up study of a vaccination programme against cutaneous leishmaniasis. II. Vaccination with a recently isolated strain of L. tropica from Jericho. Trans R Soc Trop Med Hyg. 1972;66(2):239-43. doi: 10.1016/0035-9203(72)90153-8. No abstract available. PMID 5048790
- [Background] Modabber F. Experiences with vaccines against cutaneous leishmaniasis: of men and mice. Parasitology. 1989;98 Suppl:S49-60. doi: 10.1017/s0031182000072243. PMID 2657601